CLINICAL TRIAL: NCT04764591
Title: Effect of Different Approaches of Infraclavicular Brachial Plexus Block on Tissue Perfusion: A Randomized Trial
Brief Title: Tissue Perfusion for Different Approaches of Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, assistant professor dr, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020/24-10
Record Dates: First submitted 2021-02-10; First posted 2021-02-21 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Upper Extremity Fracture; Regional Anesthesia; Brachial Plexus Blocks; Perfusion Index; Tissue Perfusion
Keywords: lateral sagittal approach; costoclavicular approach; block success; perfusion index; brachial plexus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral sagittal approach (Active Comparator): Patients in this group will be randomized to receive a lateral sagittal approach for Ultrasound Guided Infraclavicular Brachial Plexus Nerve Block .
  Interventions: Other: Lateral sagittal approach
- Costoclavicular approach (Active Comparator): Patients in this group will be randomized to receive a costoclavicular approach to Ultrasound Guided Infraclavicular Brachial Plexus Nerve Block .
  Interventions: Other: Costoclavicular approach

INTERVENTIONS:
Other: Lateral sagittal approach — Lateral sagittal approach for ultrasound guided infraclavicular brachial plexus block
  Arms: Lateral sagittal approach
Other: Costoclavicular approach — Costoclavicular approach for ultrasound guided infraclavicular brachial plexus block
  Arms: Costoclavicular approach

SUMMARY:
To compare the two different approaches of infraclavicular brachial plexus block in forearm, wrist and hand surgery in terms of perfusion index, tissue oxygenation, sensory and motor block onset time and total effect time, first analgesic time, side effects and complications, and duration of block application.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo elective forearm or hand surgery under infraclavicular brachial plexus block
* American Society of Anesthesiologists class 1 to 3
* Ability to consent

Exclusion Criteria:

* History of allergic reaction to local anaesthetics
* Peripheral neuropathy
* Renal or hepatic insufficiency
* Coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
perfusion index | up to motor block scale ≥3
  the effect of the block on the perfusion index
tissue oxygenation | up to motor block scale ≥3
  the effect of the block on the tissue oxygenation

SECONDARY OUTCOMES:
motor block onset time | Assessed 40 minutes after block completion
  quality of motor block scale ≥2
sensorial block onset time | up to 24 hours
  quality of sensorial block scale ≥2
complications | up to 24 hours
  block related complications such as pneumothorax, vascular injury, local anesthetic systemic toxicity
duration of block application | during the intervention
  from the needle puncture to the end of the local anesthetic injection

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baytar C, Koksal BG. Effects of different approaches of infraclavicular brachial plexus block on perfusion index and tissue perfusion. Ann Med. 2025 Dec;57(1):2451765. doi: 10.1080/07853890.2025.2451765. Epub 2025 Jan 11. PMID 39797918